CLINICAL TRIAL: NCT03736642
Title: Study of the Microbiological Profile of Stool in Patients With Anorexia Nervosa
Acronym: ANOSTOOL
Status: Withdrawn | Type: Observational
Why Stopped: never started
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 18CH109; 2018-A01731-54 (Other: ANSM)
Record Dates: First submitted 2018-11-02; First posted 2018-11-09 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Anorexia Nervosa; Eating Disorder
Keywords: stool; constitutional thinness
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 20 g of stool
  * 18 ml of urines
  * 12 ml of blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- restrictive anorexia nervosa with hunger
  Interventions: Biological: blood sampling; Other: stool sampling; Other: urine sampling; Diagnostic Test: neuropsychological tests
- restrictive anorexia nervosa without hunger
  Interventions: Biological: blood sampling; Other: stool sampling; Other: urine sampling; Diagnostic Test: neuropsychological tests
- constitutional thinness
  Interventions: Biological: blood sampling; Other: stool sampling; Other: urine sampling; Diagnostic Test: neuropsychological tests
- control subjects without eating disorders
  Interventions: Biological: blood sampling; Other: stool sampling; Other: urine sampling; Diagnostic Test: neuropsychological tests

INTERVENTIONS:
Biological: blood sampling — 12 ml sample
Other: stool sampling — 20 g sample
Other: urine sampling — 18 ml sample
Diagnostic Test: neuropsychological tests — * Go-nogo
  * flexibility
  * food stroop
  * implicit and explicit evaluation
  * Child Depression Inventory
  * Hamilton Depression Rating Scale

SUMMARY:
Anorexia nervosa is an eating disorder whose symptomatology induces a modification of the intestinal microbiota. To date, studies have shown variable profiles without linking them to metabolic and neuropsychological energy phenotyping. This intestinal dysbiosis could be involved in the maintenance of the disorders. Bidirectional communication channels exist between the microbiota, the intestine and the brain. Anomalies in these pathways could explain the impact of the microbiota on the pathophysiology of anorexia nervosa. Therapeutic interventions would then be possible to restore the microbiota in anorexia nervosa and influence the treatment of this disease. This study aims to explore the hypothesis of disruption of the microbiota-intestinal-brain axis transversely and measuring the intestinal microbiota, urinary metabolome, biological factors nutritional, immunological and physiological plasma plasma of the intestine, and finally, the psychological dimensions characteristic of anorexia nervosa.

ELIGIBILITY:
Inclusion criteria common to all four groups

* Patient affiliated or entitled to a social security scheme
* Patient who received informed information about the study
* Patient does not object to participating in the study

Inclusion criteria specific to mental anorexia

* BMI between 13 and 17.5 kg/m2
* Diagnostic and Statistical Manual of Mental Disorders IV restrictive anorexia nervosa diagnostic criteria
* Evolution of the troubles since less than 1 year.
* with feeling of hunger: "hunger" = total score on the 24-hour hunger scale > 15 and presence of the three prandial peaks (score = 3)
* having lost the feeling of hunger: "not hungry" = total score on the 24-hour hunger scale ≤ 5 and absence of the three prandial peaks (score ≤ 2)

Inclusion criteria specific to constitutionally thin patients

* BMI between 13 and 17.5 kg/m2
* Stable weight for at least 3 months
* No eating disorder
* No markers of undernutrition

Inclusion criteria specific to normal weight subjects

* 20 kg/m2 ≤ BMI ≤ 25 kg/m2
* Stable weight for at least 3 months
* No eating disorder
* No markers of undernutrition

Non-inclusion criteria for all subjects :

* Antibiotic treatment during the 2 months preceding the sampling.
* History of immune system/autoimmune disease: Immune deficiency, Crohn's disease, systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, psoriasis, Behçet's disease, celiac disease, type I diabetes.
* History of metabolic pathology: intestinal malabsorptive disease
* Medical or surgical history deemed by the investigator to be incompatible with this study.
* Severe progressive condition other
* Pregnant woman
* Majors under guardianship or subjects deprived of their liberty by judicial or administrative decision
* Ongoing psychotropic treatment
* Progressive diarrhea (Bristol Type V and VI)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only female
Study Population: * anorexia nervosa with and without hunger
  * constitutional leanness
  * control subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
determination of bacterial microbiological profile by 16s sequencing of stool samples | at inclusion

SECONDARY OUTCOMES:
Determination of the metabolomic profile | at inclusion
  evaluated by mass spectrometry (MS/MS) of urine
Neurocognitive evaluation | at 2 months
  evaluated with questionnaire go-nogo
Neurocognitive evaluation | at 2 months
  evaluated with questionnaire of flexibility
Neurocognitive evaluation | at 2 months
  evaluated with questionnaire : food troop
Neurocognitive evaluation | at 2 months
  evaluated with questionnaires : implicit and explicit evaluation.
Psychometric scaling for thymic evaluation | at 2 months
  evaluated with questionnaire : Child Depression Inventory
Psychometric scaling for thymic evaluation | at 2 months
  evaluated with questionnaire : Hamilton Depression Rating Scale
Determination of the plasma profile of intestinal physiology markers and immunological markers | at inclusion
  Intestinal permeability markers: ASCA, antiglycan, anti GP2 IgG/IgA, calprotectin
Determination of the plasma profile of intestinal physiology markers and immunological markers | at inclusion
  immunoglobulin repertoire: A and M, inflammatory molecules: C-reactive protein
Determination of the plasma profile of intestinal physiology markers and immunological markers | at inclusion
  circulating interleukins of the Th17 profile: IL17, IL23, IL6, IL1β, IL 22, IL21, IL33, IL31, TNFα, IFNγ, IL9, IL10, IL4.

CONTACTS AND LOCATIONS:
Overall Officials: Natacha GERMAIN, Principal Investigator — CHU de Saint Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No